CLINICAL TRIAL: NCT04396964
Title: A Natural History of Perioperative Metabolism
Status: Completed | Type: Observational
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, William G Tharp, Assistant Professor, University of Vermont Medical Center
Other Study IDs: M14-291
Record Dates: First submitted 2020-05-15; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Surgery; Anesthesia; Insulin Sensitivity; Metabolic Stress Hyperglycemia
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- surgery: subjects undergoing multilevel lumbar fusion

SUMMARY:
The process of surgery is a controlled trauma to the body. Trauma induces changes in metabolic function that have evolved to help the body survive injury. The normal balance among use of sugar, fat, and protein for energy production is thought to change during trauma and surgery. This altered metabolic function may contribute to adverse outcomes from surgical procedures especially in the setting of patients with obesity or Type 2 Diabetes Mellitus. However, very little is known about the specific changes in metabolism that occur during surgical procedures.

The main objective of this project is to describe the metabolic changes that occur during a typical surgical procedure in detail. In order to measure the alterations in the balanced use of sugar, fat, and protein during surgery we will collect blood samples from patients before, during, and after spinal surgical procedures. Subjects will be enrolled in the pre-operative hold area, give informed consent, and have a dedicated peripheral IV catheter placed. We will recruit patients who are normal weight without diabetes, obese without diabetes, and obese with diabetes. The first specific aim is to characterize the metabolic changes in sugar, fat, and protein balance during surgery in metabolically normal subjects. The second specific aim to examine if there are differences in these changes in subjects who are obese or have diabetes. The final specific aim is to measure the changes in metabolism at high resolution using a method called metabolomics, which is analogous to genome profiling. This method measures hundreds of compounds produced in different amounts as metabolic balance changes.

The major impacts that may be derived from these data range from a more thorough understanding of metabolism under trauma to identification of new markers for risk stratification and intervention to improve clinical outcomes. These data will help build the foundation for new approaches to understanding the physiological and metabolic responses to stress and trauma.

DETAILED DESCRIPTION:
We will conduct a cross-sectional study in a cohort of patients undergoing spinal surgery for discectomy, laminectomy, or vertebral fixation. We will recruit a cohort of subjects in groups with metabolic phenotypes defined by body mass index (BMI) and glycemic control. We are choosing to use spinal surgeries as they utilize inhaled anesthetics, run hours in length, do not involve ischemic tourniquet time, and use basic elements of the anesthetic pharmacopeia including anti-emetics, opioid analgesics, and paralytics. Further the increased surgical stress of entering the thorax or peritoneum are avoided. These features provide a long steady-state of surgical intervention with minimal additional maneuvers allowing for a controlled examination of surgical metabolism.

The categorical criteria for the groups will be body type: lean (BMI<25), overweight (BMI >25, <30), and obese (BMI >30 but <40), and glycemia: normoglycemic (fasting blood glucose; FBG <100 mg/dL or HbA1c <5.5%), impaired fasting glucose (FBG >100 mg/dL and <126 mg/dL, or HbA1c >5.5% and <6.5%), Type 2 Diabetes (FBG >126 mg/dL or HbA1c >6.5%).

Subjects will be screened, enrolled, give informed consent, and have a dedicated peripheral IV line placed in pre-operative hold. A baseline blood sample will be collected in pre-operative hold, after transfer to the table in the operating room, and immediately prior to induction of anesthesia. Following induction blood samples will be collected at 15' intervals for the initial 2 hours of each case, then at 30' intervals for the remainder of the case and for 2 hours in the post-anesthesia care unit. Samples will be processed and stored at -80C until analyzed. Intra-operative data from the anesthesia record will be collected and included in the study database.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were eligible if they were >18 years old without acute or chronic health conditions who were undergoing multilevel lumbar fusions with an inhaled anesthetic.

Exclusion Criteria:

* acute or chronic health conditions including cardiac, pulmonary, hepatic, renal, auto-immune, or hematological disease. Obese subjects with body mass index >40kg/m2 were excluded. Subjects with Type 2 diabetes were eligible if they were well-controlled (HbA1c <7.5%) and treated with diet and exercise, metformin, or insulin. Subjects were excluded if taking a sulfonylurea, thiazolidindiones, DPP-4 inhibitor, GLP-1 analog, weight loss medication, or other medications affecting glucose homeostasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing multilevel lumbar fusion with an inhaled anesthetic.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2016-11-03 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
glucose | perioperative
  glucose concentrations
insulin | perioperative
  insulin concentrations
c-peptide | perioperative
  c-peptide concentrations
cortisol | perioperative
  cortisol concentrations

IPD SHARING:
Plan to Share IPD: No